CLINICAL TRIAL: NCT07370779
Title: The Effect Of Positive End-Expiratory Pressure on Optic Nerve Sheath Diameter In Pediatric Patients Undergoing Craniotomy in Supine Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eren Karahan, Md, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LutfiKırdarCityHospital
Record Dates: First submitted 2025-12-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Craniotomy Surgery; Pediatric Patient Safety; Pediatric Patient; Positive End-expiratory Pressure (PEEP); Optic Nerve Sheath Diameter Measurement
Keywords: peep; pediatric patients; optic nerve sheath diameter; intracranial pressure; craniotomy
MeSH Terms: interventions — Anesthesia, General; Anesthetics; Respiration, Artificial

STUDY DESIGN:
Intervention Model Description: The initial group (Study Group) received a PEEP level of 4 cmH2O. Tthe second group (Control Group) received no PEEP.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): PEEP 4 group
  Interventions: Drug: General Anesthesia; Drug: Anesthetic Agents; Device: mechanical ventilation (MV)
- Control Group (Active Comparator): PEEP 0 Group
  Interventions: Drug: General Anesthesia; Drug: Anesthetic Agents; Device: mechanical ventilation (MV)

INTERVENTIONS:
Drug: General Anesthesia — General anesthesia was administered according to standard clinical practice, including intravenous induction agents and inhalational anesthetics, as part of routine perioperative care.
Drug: Anesthetic Agents — Anesthetic agents, including propofol, fentanyl, rocuronium, and sevoflurane, were used as part of standard anesthetic management during the procedure.
Device: mechanical ventilation (MV) — Mechanical ventilation was provided using a standard anesthesia ventilator in volume-controlled mode during surgery.

SUMMARY:
This study evaluated the effect of positive end-expiratory pressure (PEEP) on optic nerve sheath diameter (ONSD), an indicator of intracranial pressure, in pediatric patients undergoing craniotomy in the supine position. The findings indicated that the application of PEEP did not result in a significant difference in ONSD. Although a significant decrease in systolic and diastolic blood pressure was observed with the use of PEEP, these values remained within normal ranges and did not indicate adverse hemodynamic effects. The results suggest that the use of a PEEP level of 4 cmH2O in pediatric patients with intracranial masses is safe and may be applied during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 6 months to 18 years
* American Society of Anesthesiologists (ASA) physical status III
* Scheduled for elective craniotomy in the supine position
* Presence of an extra-axial intracranial mass
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Open fontanelles
* Orbital pathology
* Severe increases in intracranial pressure associated with nausea, vomiting, visual disturbances, or seizures
* Radiologic or clinical signs of brain herniation
* Hydrocephalus
* Cerebral infection
* Congenital syndromes
* History of surgery involving the optic nerve
* Use of inotropic therapy
* Hemodynamic instability
* Surgical complications during the operation or procedures lasting longer than 8 hours
* Postoperative intubation requiring intensive care unit follow-up
* Tumors invading the optic nerve
* Inability to obtain written informed consent from parents or legal guardians

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter | Four times in during the operation by using ultrasonography. T0: before induction of anesthesia; T1: immediately after the dura was opened; T2: just before the dura was closed; T3: before extubation

SECONDARY OUTCOMES:
Heart Rate | Four times in during the operation. T0: before induction of anesthesia; T1: immediately after the dura was opened; T2: just before the dura was closed; T3: before extubation
systolic blood pressure | Four times in during the operation. T0: before induction of anesthesia; T1: immediately after the dura was opened; T2: just before the dura was closed; T3: before extubation
diastolic blood pressure | Four times in during the operation. T0: before induction of anesthesia; T1: immediately after the dura was opened; T2: just before the dura was closed; T3: before extubation
Peripheral oxygen saturation | Four times in during the operation. T0: before induction of anesthesia; T1: immediately after the dura was opened; T2: just before the dura was closed; T3: before extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Lutfi Kırdar City Hospital, Istanbul, eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sezen O, Saracoglu KT, Simsek T, Cevik B, Aydogmus E. The effect of positive end-expiratory pressure on optic nerve diameter in patients undergoing craniotomy operation. Ann Clin Anal Med. 2021;12(02):199-203.
- [Background] Pulitano S, Mancino A, Pietrini D, Piastra M, De Rosa S, Tosi F, De Luca D, Conti G. Effects of positive end expiratory pressure (PEEP) on intracranial and cerebral perfusion pressure in pediatric neurosurgical patients. J Neurosurg Anesthesiol. 2013 Jul;25(3):330-4. doi: 10.1097/ANA.0b013e31828bac4d. PMID 23519374
- [Background] Padayachy L, Brekken R, Fieggen G, Selbekk T. Noninvasive Transorbital Assessment of the Optic Nerve Sheath in Children: Relationship Between Optic Nerve Sheath Diameter, Deformability Index, and Intracranial Pressure. Oper Neurosurg. 2019 Jun 1;16(6):726-733. doi: 10.1093/ons/opy231. PMID 30169680
- [Background] Khandelwal A, Kapoor I, Mahajan C, Prabhakar H. Effect of Positive End-Expiratory Pressure on Optic Nerve Sheath Diameter in Pediatric Patients with Traumatic Brain Injury. J Pediatr Neurosci. 2018 Apr-Jun;13(2):165-169. doi: 10.4103/jpn.JPN_112_17. PMID 30090129